CLINICAL TRIAL: NCT03196180
Title: A Feasibility Trial of Alternating Intravaginal Application of 5-Fluorouracil and Imiquimod for Treatment of High-Grade Cervical Squamous Intraepithelial Lesions
Brief Title: Topical Fluorouracil and Imiquimod in Treating Patients With High-Grade Cervical Intraepithelial Neoplasia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2017-01079; NCI-2017-01079 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); N01-CN-2012-00031; 1712088061 (Other: University of Arizona Cancer Center - Prevention Research Clinic); UAZ2016-08-02 (Other: DCP); N01CN00031 (NIH); P30CA023074 (NIH)
Record Dates: First submitted 2017-06-21; First posted 2017-06-22 (Actual); Results first posted 2022-02-23 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Cervical Intraepithelial Neoplasia Grade 2/3; Cervical Squamous Cell Carcinoma In Situ; Cervical Squamous Intraepithelial Neoplasia 2; High Grade Cervical Intraepithelial Neoplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — Imiquimod; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (topical fluorouracil, imiquimod) (Experimental): Patients receive topical fluorouracil intravaginally via applicator at weeks 1, 3, 5, 7, 9, 11, 13, and 15 and imiquimod intravaginally via applicator at weeks 2, 4, 6, 8, 10, 12, 14, and 16. Patients who are menstruating will delay application until the end of the menstrual cycle.
  Interventions: Drug: Imiquimod; Drug: Topical Fluorouracil

INTERVENTIONS:
Drug: Imiquimod — Given intravaginally
  Other Names: Aldara; R 837; S 26308; Zyclara
Drug: Topical Fluorouracil — Given intravaginally
  Other Names: Actino-Hermal; Arumel; Carac; Cytosafe; Efudex; Efurix; Fiverocil; Fluoroplex; Flurox; Timazin; Tolak

SUMMARY:
This early phase I clinical trial studies the side effects of topical fluorouracil and imiquimod ointment in treating patients with high-grade cervical intraepithelial neoplasia. Topical fluorouracil may kill precancerous cells. Imiquimod ointment may stimulate the immune system. Applying topical fluorouracil and imiquimod ointment may cause fewer side effects and may be a better way to treat patients with precancerous cervical lesions.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Assess feasibility, evaluated based on safety and tolerability, of a combination agent intervention (once-weekly self-administered intravaginal application of 5-fluorouracil alternating with once-weekly provider-applied imiquimod) for treatment of high-grade cervical squamous intraepithelial lesions.

SECONDARY OBJECTIVES:

I. Assess efficacy of the combination agent intervention on cervical disease regression (endpoint based on histologic regression from high-grade lesions to low-grade or no lesions and clearance of high risk-human papillomavirus [HPV] detection) between baseline and study exit visits.

II. Assess efficacy of the combination agent intervention on genotype-specific HPV clearance between baseline and study exit visits.

III. Assess efficacy of the combination agent intervention on biomarkers of local immune activation (measurement of changes in expression of Toll-like receptors (TLR) and T-regulatory cells and the levels of innate, immune mediating and proinflammatory cytokines with intravaginal 5-fluorouracil [FU] and imiquimod) between baseline and study exit visits.

OUTLINE: This is a phase I, dose escalation study of imiquimod.

Patients receive topical fluorouracil intravaginally via applicator at weeks 1, 3, 5, 7, 9, 11, 13, and 15 and imiquimod intravaginally via applicator at weeks 2, 4, 6, 8, 10, 12, 14, and 16. Patients who are menstruating will delay application until the end of the menstrual cycle.

After completion of study treatment, patients are followed up within 8 months.

ELIGIBILITY:
Inclusion Criteria:

* Women with biopsy confirmed high grade cervical squamous intraepithelial lesions (i.e., cervical squamous intraepithelial neoplasia 3 [CIN3] lesions, and cervical squamous epithelial neoplasia 2 [CIN2] lesions with diagnosis confirmed by positive p16 immunohistochemistry staining) within 12 weeks of baseline visit
* Karnofsky >= 70%
* Leukocytes >= 3,000/microliter
* Absolute neutrophil count >= 1,500/microliter
* Platelets >= 100,000/microliter
* Serum creatinine =< the upper institutional limits
* Participants must have a negative human immunodeficiency virus (HIV) antibody/antigen test and negative Chlamydia (C.) trachomatis/Neisseria (N.) gonorrhea nucleic acid amplification test (NAAT)
* Agree to use an effective form of contraception; the effects of intravaginal 5-fluorocuracil and imiquimod on the developing human fetus at the recommended therapeutic dose are unknown; for this reason and because 5- fluorouracil is known to be teratogenic, women of child-bearing potential must agree to use adequate dual methods of contraception (hormonal method of birth control, intrauterine device, or tubal ligation - plus condoms) or abstinence prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Women treated previously with 5-fluorouracil or imiquimod or other medications for high-grade squamous intraepithelial lesions will be excluded from the study
* Concurrent vaginal, vulvar, anal lesions or symptomatic infections
* Pregnant or planning pregnancy within the next 6 months, or breastfeeding; pregnant women are excluded from this study because 5-fluorouracil is an antimetabolite with the potential for teratogenic effects; because there is an unknown but potential risk for adverse events (AEs) in nursing infants secondary to treatment of the mother with 5-fluorouracil, breastfeeding should be discontinued if the mother is treated with 5-fluorouracil
* Inability to speak or read English or Spanish
* Prior hysterectomy
* Use of anticoagulant medications
* Subjects who have a known immunocompromised condition (HIV positive [+], use of immunosuppressive medications or systemic steroids, organ transplant recipients) or autoimmune conditions (e.g. psoriasis, rheumatoid arthritis or other known autoimmune conditions)
* Evidence of invasive anal, vulva, vaginal, or cervical carcinoma; prior loop electrosurgical excision procedure (LEEP) or ablative treatment within 6 months prior to study entry; other invasive malignancies, with the exception of non-melanoma skin cancer, within the last 5 years
* Pathologic findings consistent with

  * Atypical endometrial cells or serious glandular-cell atypia (atypical glandular cells, favor neoplasia cytology diagnosis)
  * Evidence of cervical carcinoma on Pap smear or biopsy
  * More than two cervical quadrants of CIN 3 as visualized by colposcopy
  * Nonvisual squamous columnar junction on colposcopy with no concurrent endocervical sampling performed
* Use of other investigational agents within 6 months prior to enrollment
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to 5-fluorouracil or imiquimod
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection (other than human papilloma virus [HPV]), symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Subjects with known partial or complete dihydropyrimidine dehydrogenase (DPD) enzyme deficiency

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-11-04 (Actual); Study Completion 2024-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Rahangdale, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Topical Fluorouracil, Imiquimod): Patients receive once-weekly intravaginal application of 5-fluorouracil and imiquimod used on alternating weeks for 8 to 16 weeks.
  Imiquimod: Given intravaginally
  Topical Fluorouracil: Given intravaginally
Period: Overall Study
Arm/Group | Treatment (Topical Fluorouracil, Imiquimod)
Started | 13
Completed | 11
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Topical Fluorouracil, Imiquimod)
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 27 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 7
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Intravaginal Use 5-FU and Imiquimod on Alternating Weeks in Women With Biopsy Confirmed High Grade Cervical Squamous Intraepithelial Lesions.
Description: Feasibility is evaluated based on safety and tolerability of the study intervention. For safety, the study assessed the number of participants experiencing the specified adverse events defined as Grade 2 or greater toxicity (or Grade 1 toxicity of any genital lesion (blisters, ulcerations, or pustules)) that is possibly, probably, or definitely related and lasts for more than 5 days. For tolerability, the study assessed the number of participants who were not able to apply at least 50% of the treatment due to the specified adverse events.
Time Frame: Up to 22 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Topical Fluorouracil, Imiquimod)
Number analyzed (Participants) | 13
Participants
  Safety | 4
  Tolerability | 1

2. Secondary Outcome: Response to Intravaginal 5-FU and Imiquimod Defined as Histologic Regression and Clearance of High-risk Human Papilloma Virus (HR-HPV)
Description: The response will be reported along with their 95% confidence intervals. Response is defined as histologic regression from high-grade lesions to low-grade- or no lesions and clearance of HR-HPV detection between baseline and end of study.
Time Frame: At end of study visit (4-6 weeks after the last agent application)
Population: Participants who were HR-HPV negative at baseline were excluded from the analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Topical Fluorouracil, Imiquimod)
Number analyzed (Participants) | 10
percentage of participants | 40 [12 to 74]

3. Secondary Outcome: Type Specific Human Papillomavirus (HPV) Clearance
Description: The type-specific HR-HPV clearance will be reported along with their 95% confidence intervals.
Time Frame: At end of study visit (4-6 weeks after the last agent application)
Population: Participants positive for a given HPV genotype at baseline were assessed for the clearance of this genotype at the end of study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Topical Fluorouracil, Imiquimod)
Number analyzed (Participants) | 12
percentage of participants
  HPV16: number analyzed (Participants) | 4
  HPV16 | 75 [19 to 99]
  HPV31: number analyzed (Participants) | 2
  HPV31 | 50 [1 to 99]
  HPV35: number analyzed (Participants) | 1
  HPV35 | 100 [3 to 100]
  HPV39: number analyzed (Participants) | 1
  HPV39 | 0 [0 to 98]
  HPV51: number analyzed (Participants) | 2
  HPV51 | 0 [0 to 84]
  HPV52: number analyzed (Participants) | 4
  HPV52 | 75 [19 to 99]
  HPV56: number analyzed (Participants) | 1
  HPV56 | 0 [0 to 98]
  HPV66: number analyzed (Participants) | 2
  HPV66 | 50 [1 to 99]
  HPV68: number analyzed (Participants) | 2
  HPV68 | 100 [16 to 100]

4. Secondary Outcome: Change in Expression of Biomarkers of Local Immune Activation (Cytokines) After Treatment With Self-administered Intravaginal Topical Fluorouracil and Imiquimod
Description: For each biomarker, the mean change of log transformed data and the associated standard deviation will be reported. Will measure the innate (IFN-alpha2), immune mediating (IFN-gamma, IL-10, IL-12), and pro-inflammatory (IL-1alpha, -1beta, -6, -8, MIP-1alpha, TNF) cytokine.
Time Frame: Baseline to up to end of study visit (4-6 weeks after last agent application)
Population: Participants with data at both baseline and end of study for a given biomarker were included in the analysis.
Measure: Mean (Standard Deviation); unit: log pg/ml
Arm/Group | Treatment (Topical Fluorouracil, Imiquimod)
Number analyzed (Participants) | 12
log pg/ml
  IFN-alpha 2: number analyzed (Participants) | 10
  IFN-alpha 2 | -0.29 (1.49)
  IFN-gamma: number analyzed (Participants) | 9
  IFN-gamma | 0.16 (0.81)
  IL-1 alpha: number analyzed (Participants) | 11
  IL-1 alpha | -0.55 (1.01)
  IL-1 beta: number analyzed (Participants) | 10
  IL-1 beta | -0.15 (1.84)
  IL-6: number analyzed (Participants) | 11
  IL-6 | -0.84 (1.94)
  IL-8: number analyzed (Participants) | 11
  IL-8 | -0.16 (2.63)
  IL-12: number analyzed (Participants) | 9
  IL-12 | 0.15 (0.95)
  IL-13: number analyzed (Participants) | 10
  IL-13 | -0.53 (1.11)
  MIP-1 alpha: number analyzed (Participants) | 6
  MIP-1 alpha | 0.66 (0.77)
  TNF alpha: number analyzed (Participants) | 9
  TNF alpha | -0.01 (1.99)

5. Secondary Outcome: Change in Expression of Biomarkers of Local Immune Activation (Toll Like Receptors (TLRs)) After Treatment With Self-administered Intravaginal Topical Fluorouracil and Imiquimod
Description: For each biomarker, the mean change of log transformed data and the associated standard deviation will be reported. TLR messenger ribonucleic acid expression is normalized by the housekeeping genes and does not have a unit of measure.
Time Frame: Baseline to up to end of study visit (4-6 weeks after last agent application)
Population: Participants with data at both baseline and end of study for a given biomarker were included in the analysis.
Measure: Mean (Standard Deviation); unit: gene expression level
Arm/Group | Treatment (Topical Fluorouracil, Imiquimod)
Number analyzed (Participants) | 12
gene expression level
  TLR2: number analyzed (Participants) | 11
  TLR2 | 0.90 (2.16)
  TLR3 | 0.75 (4.26)
  TLR4: number analyzed (Participants) | 10
  TLR4 | 0.86 (1.84)
  TLR7: number analyzed (Participants) | 10
  TLR7 | 2.20 (1.36)
  TLR9 | 0.95 (4.43)

ADVERSE EVENTS:
Time Frame: 14-22 weeks
Arm/Group | Treatment (Topical Fluorouracil, Imiquimod)
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 13/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Topical Fluorouracil, Imiquimod) (N=13)
Abdominal pain (Gastrointestinal disorders) | 1
Pain - Lower abdominal (Gastrointestinal disorders) | 2
Fever (General disorders) | 1
Flu like symptoms (General disorders) | 1
Other (General disorders) | 2
Bacterial vaginosis (Infections and infestations) | 1
Candida (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 5
Weight gain (Investigations) | 3
Weight loss (Investigations) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 4
Dysuria (Renal and urinary disorders) | 1
Cervical erythema (Reproductive system and breast disorders) | 1
Cervical friability (Reproductive system and breast disorders) | 1
Dysmenorrhea/cramping with menses (Reproductive system and breast disorders) | 2
Dyspareunia (Reproductive system and breast disorders) | 1
Metrorrhagia (Reproductive system and breast disorders) | 1
Pain - Pelvic (Reproductive system and breast disorders) | 6
Pain - Vagina (Reproductive system and breast disorders) | 8
Postcoital bleeding (Reproductive system and breast disorders) | 1
Unexplained infrequent bleeding (Reproductive system and breast disorders) | 4
Vaginal abrasions (Reproductive system and breast disorders) | 1
Vaginal discharge as observed by clinician (Reproductive system and breast disorders) | 1
Vaginal erythema (Reproductive system and breast disorders) | 1
Vaginal discharge by participant report (Reproductive system and breast disorders) | 7
Vaginal lesions (Reproductive system and breast disorders) | 3
Vulvar/vaginal itching (Reproductive system and breast disorders) | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Hypertension (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-04): https://cdn.clinicaltrials.gov/large-docs/80/NCT03196180/Prot_SAP_000.pdf